CLINICAL TRIAL: NCT06336850
Title: Safety and Efficacy of Endoscopic Ultrasound-Guided Portal Pressure Gradient Measurement
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 069.GID.2020.D
Record Dates: First submitted 2021-12-09; First posted 2024-03-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Liver Diseases
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Patients undergoing Endoscopic-Ultrasound Guided liver biopsies and Endoscopic Ultrasound-Guided Portal Pressure Gradient Measurements
  Interventions: Procedure: Endoscopic Ultrasound-Guided Portal Pressure Gradient Measurement

INTERVENTIONS:
Procedure: Endoscopic Ultrasound-Guided Portal Pressure Gradient Measurement — The endoscopic ultrasound (EUS)-guided 25G fine needle aspirate (FNA) needle procedure is a straightforward minimally invasive technique for direct portal pressure measurements.

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, and adequacy of Endoscopic Ultrasound (EUS) Portal Pressure Gradient Measurement (PPGM) in patients undergoing EUS-guided liver biopsies.

DETAILED DESCRIPTION:
Patients undergoing EUS-guided liver biopsy may qualify to participate in this study. The purpose of this study is to evaluate the efficacy, safety, and adequacy of EUS- Portal Pressure Gradient Measurement (PPGM) in patients with liver disease referred for EUS-guided liver biopsy.

ELIGIBILITY:
INCLUSION CRITERIA

* Age 18 years or older
* Patient who has been referred for EUS procedure and direct PPG measurement and -undergoing EUS-guided liver biopsy
* History of liver disease or suspected cirrhosis and considered for PPGM

EXCLUSION CRITERIA

* Patient is less than 18 or greater than 85 years of age
* Patient is pregnant, breast-feeding, or planning to become pregnant during the course of the study
* Patient is unwilling or unable to sign and date the informed consent
* Patient for whom endoscopic procedures are contraindicated.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-12-23 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Portal Pressure Gradient Measurements from Hepatic and Portal Veins | 2 years
  A catheter is inserted into the hepatic vein before hepatic venous pressure and portal vein pressure are recorded

SECONDARY OUTCOMES:
Correlation between Portal Pressure Gradient Measurements and the presence or absence of portal hypertension | 2 years
  Statistical tests to determine relationship between portal pressure gradient measurements and portal hypertension
Clinical significance between portal pressure gradient measurement and portal hypertension | 2 years
  Presence of varices, hypertensive gastropathy, or thrombocytopenia.

CONTACTS AND LOCATIONS:
Overall Officials: Prashant Kedia, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States